CLINICAL TRIAL: NCT07173907
Title: Comparison of Epithelium-on CuRV and Epithelium-off aCXL Protocols in the Management of Keratoconus
Brief Title: Epi-on CuRV and Epi-off aCXL Protocols in the Management of Keratoconus
Acronym: CuRVaCXL
Status: Completed | Type: Observational
Sponsor: Gemini Eye Clinic (Industry)
Responsible Party: Principal Investigator, Dr. Pavel Stodulka, Principal Investigator, Gemini Eye Clinic
Other Study IDs: CXL2025; 2019-18 (Other: Gemini Eye Clinics)
Record Dates: First submitted 2025-09-08; First posted 2025-09-15 (Actual); Last update posted 2025-09-15 (Actual); Status verified 2025-08

CONDITIONS: Keratoconus
MeSH Terms: conditions — Keratoconus

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- CuRV CXL protocol cohort: The subjects underwent the procedure of CuRV method that was performed as an outpatient procedure under topical anesthesia (tetracaine 1%). A two-part transepithelial isotonic riboflavin system (ParaCel™ Part 1 and Part 2) was used. Part 1 was applied with a surgical spear and repeated drops, followed by Part 2 instillation for 6 minutes. After rinsing with balanced salt solution, UVA irradiation was performed using the Mosaic® device with Boost Goggles™ delivering supplemental oxygen. Pulsed UVA (365 nm, 30 mW/cm²) was applied in a personalized, three-zone pattern (15 J/cm² to the cone apex, 10 J/cm² to an intermediate annulus, and 7.2 J/cm² to the periphery), guided by Pentacam tomography. A bandage contact lens was placed at the end of the procedure.
  Interventions: Procedure: CuRV CXL
- Accelerated CXL Procedure (aCXL): The subjects underwent the aCXL procedure was performed under topical anesthesia after tailored epithelial removal, leaving a small island over the thinnest corneal area. Riboflavin-dextran solution was applied for 30 minutes, followed by UVA irradiation (9 mW/cm², total 5.4 J/cm²) using the KXL device. The cornea was rinsed with Ringer's solution during treatment, and a bandage contact lens was placed afterward.
  Interventions: Procedure: Accelerated CXL Procedure (aCXL)

INTERVENTIONS:
Procedure: CuRV CXL — A two-part transepithelial isotonic riboflavin system (ParaCel™ Part 1 and Part 2) was used. Part 1 was applied with a surgical spear and repeated drops, followed by Part 2 instillation for 6 minutes. After rinsing with balanced salt solution, UVA irradiation was performed using the Mosaic® device with Boost Goggles™ delivering supplemental oxygen. Pulsed UVA (365 nm, 30 mW/cm²) was applied in a personalized, three-zone pattern (15 J/cm² to the cone apex, 10 J/cm² to an intermediate annulus, and 7.2 J/cm² to the periphery), guided by Pentacam tomography. A bandage contact lens was placed at the end of the procedure.
  Groups: CuRV CXL protocol cohort
Procedure: Accelerated CXL Procedure (aCXL) — The subjects underwent the aCXL procedure was performed under topical anesthesia after tailored epithelial removal, leaving a small island over the thinnest corneal area. Riboflavin-dextran solution was applied for 30 minutes, followed by UVA irradiation (9 mW/cm², total 5.4 J/cm²) using the KXL device. The cornea was rinsed with Ringer's solution during treatment, and a bandage contact lens was placed afterward.
  Groups: Accelerated CXL Procedure (aCXL)

SUMMARY:
This study investigates the effectiveness and safety of two different corneal cross-linking (CXL) protocols for the management of progressive keratoconus: the accelerated epithelium-off technique (aCXL) and the topography-guided epithelium-on Customized Remodeled Vision (CuRV) protocol. These methods differ in their mode of ultraviolet-A (UVA) energy delivery and their approach to corneal surface preservation, with potential implications for both structural stabilization and patient comfort. The primary aim was to evaluate changes in corrected distance visual acuity (CDVA) and maximum keratometry (Kmax) over a 24-month follow-up period, allowing for a direct comparison of visual and topographic outcomes between the two approaches.

By assessing these endpoints, the study seeks to address whether epithelium-on, customized cross-linking can achieve similar or improved results compared with conventional accelerated epithelium-off treatment. The findings are intended to provide insights into the relative benefits of standardized versus individualized cross-linking techniques, with the broader goal of optimizing treatment strategies for patients with keratoconus.

ELIGIBILITY:
Inclusion Criteria:

* adult eyes
* progressive keratoconus (grades 1 to 3-4, Krumeich-Amsler classification)
* corneal thickness ≥400 μm
* endothelial cell density ≥1500 cells/mm²

Exclusion Criteria:

* prior corneal surgeries
* corneal scars
* dystrophies
* marginal pellucid degeneration
* systemic connective tissue disorders
* uncontrolled diabetes
* pregnancy, or breastfeeding.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with keratoconus grades 1 to 3-4 undergoing corneal cross-linking (CXL) treatment as part of routine clinical care.
Sampling Method: Non-Probability Sample
Enrollment: 135 (Actual)
Dates: Start 2016-01-01 (Actual); Primary Completion 2023-12-31 (Actual); Study Completion 2024-03-30 (Actual)

PRIMARY OUTCOMES:
Change in Maximal Corneal Curvature Keratometry Kmax | Baseline, 1 Month, 6 Months, 1 Year, 2 Years
  The difference in Kmax values measured between baseline and subsequent follow-up visits

SECONDARY OUTCOMES:
Change in Manifest refraction Spherical Equivalent | Baseline, 1 Month, 6 Months, 1 Year, 2 Years
  Change in Manifest refraction Spherical Equivalent between baseline and the subsequent follow-up.
Change in Uncorrected Distance Visual Acuity | Baseline, 1 Month, 6 Months, 1 Year, 2 Years
  Change in Uncorrected Distance Visual Acuity expressed in logMAR between baseline and the subsequent follow-up.
Change in Mean Corneal Curvature Keratometry Kmean | Baseline, 1 Month, 6 Months, 1 Year, 2 Years
  The difference in Kmean values measured between baseline and subsequent follow-up visits
Change in Corrected Distance Visual Acuity | Baseline, 1 Month, 6 Months, 1 Year, 2 Years
  Change in Corrected Distance Visual Acuity expressed in logMAR between baseline and the subsequent follow-up.
Change in Thinnest Corneal Thickness | Baseline, 1 Month, 6 Months, 1 Year, 2 Years
  The difference in thinnest corneal thickness between baseline and subsequent follow-up visits